CLINICAL TRIAL: NCT03255902
Title: Family Routine - Healthy Families
Brief Title: Family Routines - Healthy Families
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Corewell Health East (Other)
Collaborators: University of Michigan (Other)
Responsible Party: Principal Investigator, Donna Marvicsin, Nurse Practitioner, Pediatric Endocrinology, Corewell Health East
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2016-154
Record Dates: First submitted 2017-08-16; First posted 2017-08-21 (Actual); Results first posted 2019-07-26 (Actual); Last update posted 2019-07-26 (Actual); Status verified 2019-05

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: This feasibility study will be a mixed methods non-randomized trial to examine the feasibility of combining a parent skill training intervention with a family evening routine intervention. Evidence of feasibility will include attendance, activities completed, and interviews.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Families attending parenting classes (Experimental): Families attended 6 parenting sessions, filled out daily glucose screens, & questionnaires
  Interventions: Behavioral: Parenting classes

INTERVENTIONS:
Behavioral: Parenting classes — Parenting Classes:The Incredible Years curriculum

SUMMARY:
The purpose of the proposed study, Family Routines - Healthy Families, is to examine the feasibility and acceptability of a parenting/family routine intervention program for parents of young children, ages 2-5, with type 1 diabetes.

DETAILED DESCRIPTION:
The intervention in Family Routines - Healthy Families contains an established and effective parent skills training curriculum called "The Incredible Years," uniquely integrated with a newly developed family evening routine component e.g., family dinner time and evening routine, to promote improved metabolic control. The investigator will assess outcomes during and at one week post intervention. Outcome measures will include family routine, specifically the time between the dinner and bedtime glucose check, parent bedtime decision making, and child overnight glucose control. In addition, parental quality of life and receptiveness to the intervention will be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Self identification as primary care giver of child that fits following criteria:

   1. Age 2 - 5 years
   2. Diagnosis of Type 1 diabetes
   3. Most recent Hemoglobin A1c (HbA1c) > 8.0
   4. Child a patient of Pediatric Endocrinology, Beaumont Children's Hospital
2. English fluency

Exclusion Criteria:

1. Cognitively impaired
2. Does not meet inclusion criteria

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 7 (Actual)
Dates: Start 2016-05-24 (Actual); Primary Completion 2017-03-01 (Actual); Study Completion 2019-01-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donna Marvicsin, PhD, Principal Investigator — William Beaumont Children's Hospital

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Families Attending Parenting Classes
Started | 7
Completed | 5
Not Completed | 2

BASELINE CHARACTERISTICS:
Population: 7 parents enrolled with children between the ages of 2 to 5 years old, but 2 did not complete.
Arm/Group | Families Attending Parenting Classes
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Effect of Intervention on Evening Glucose Control.
Description: Number of families whose child achieved a decrease overnight between bedtime blood glucose level and morning fasting glucose level following intervention at 6 weeks.
Time Frame: After 6 weeks of classes
Population: 2 participants did not complete study
Measure: Count of Participants; unit: Participants
Arm/Group | Families Attending Parenting Classes
Number analyzed (Participants) | 5
Participants | 2

2. Secondary Outcome: Difference Between Child's Pre-intervention and 3 Month Hemoglobin A1c Value
Description: 3-month Hemoglobin A1c value subtracted from pre-intervention Hemoglobin A1c value. Positive numbers indicate an improvement in glucose control with intervention, and negative numbers indicate no improvement in glucose control with intervention.
Time Frame: Pre intervention to 3 months post intervention
Population: 2 participants did not complete study
Measure: Median (Full Range); unit: percent of HbA1c
Arm/Group | Families Attending Parenting Classes
Number analyzed (Participants) | 5
percent of HbA1c | -0.3 [-1.1 to 0.6]

ADVERSE EVENTS:
Time Frame: 6 weeks
Description: A questionnaire and survey was used to collect information for this study. Participants were carefully observed for any signs of anxiety or discomfort or any serious adverse events.
Groups:
- Families Attending Parenting Class: Families attended 6 parenting sessions, filled out daily glucose screens, & questionnaires.
  Parenting Classes: The Incredible Years curriculum
Arm/Group | Families Attending Parenting Class
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-29): https://cdn.clinicaltrials.gov/large-docs/02/NCT03255902/Prot_SAP_000.pdf